CLINICAL TRIAL: NCT05223959
Title: Culturally Adapted Psychoeducation for Bipolar Disorder in a Low-resource Setting: A Randomized Controlled Trial
Acronym: CaPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-CaPE-002
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaPE Intervention (Experimental): CaPE is a manualized intervention consisting of 12 one-to-one psychoeducation sessions, one session per week. Each session will last for 60 minutes. All sessions will be delivered by a trained therapist who will receive two months training from senior therapists before starting intervention.
  Interventions: Behavioral: Culturally adapted Psychoeducation
- Treatment as Usual (No Intervention): Treatment as usual (TAU) will be ascertained by the participant's treating physician. Research staff will record the nature and intensity of TAU delivered to each participant over a period of 3 months.

INTERVENTIONS:
Behavioral: Culturally adapted Psychoeducation — This is a culturally adapted psychoeducation program consisting of 12 sessions. Each CaPE session lasts for approximately 60 minutes, beginning with a 20-30-minute presentation on the topic of the day, followed by a related exercise (e.g., drawing a life chart or compiling a list of potential triggers for recurrence).
  Arms: CaPE Intervention

SUMMARY:
Study objectives:

1. To determine the effectiveness of the CaPE intervention compared to treatment as usual (TAU) in reducing the time to recurrence for people with bipolar disorder (BD) I/II, currently in remission in Pakistan
2. To determine the impact of the CaPE intervention compared to TAU on clinical outcomes, quality of life and functioning; and
3. To estimate the cost-effectiveness of CaPE in a low-resource setting (i.e., Pakistan) (if the RCT confirms the effectiveness of CaPE in BD.

Study design and setting:

This will be a multi-centre, assessor blind, individual, parallel-arm randomized controlled trial (RCT) with Pakistani patients with BD.

Sample Size:

The study aims to recruit a total of N=300 participants in total.

DETAILED DESCRIPTION:
Psychoeducation (PE) is an effective adjunctive treatment option in BD, however, despite the clear benefits, there are only limited, underpowered studies of PE from LMICs, including Pakistan. Therefore, the current study aims to test the effectiveness of Culturally adapted PsychoEducation (CaPE) intervention for people with BD in Pakistan. The study will include a total of N=300 people with BD from psychiatric units of teaching and non-teaching hospitals in 8 centres across Pakistan including Karachi, Lahore, Multan, Rawalpindi, Peshawar, Hyderabad, Shaheed Benazirabad and Quetta. Consented participants meeting eligibility criteria will be randomised in a 1:1 allocation to CaPE or TAU. Randomization will be computer generated and use a random permuted block method with variable block sizes stratified by site, bipolar type (I or II) and self-reported sex. Participants in CaPE intervention group will receive 12-weekly one-to-one psychoeducation sessions. Each CaPE session will last for approximately 1 hour, beginning with a 20-30-minute presentation on the topic of the day, followed by a related exercise (e.g., drawing a life chart or compiling a list of potential triggers for recurrence). Sessions will be delivered by trained psychologists who will receive regular weekly supervision to maintain fidelity. The other group will receive TAU/control group. Assessments will be carried out at baseline, months 3, 6, and 12 either in-person and/or via secure videoconference software (alternatives to in-person for COVID-19 or travel restrictions) by trained, blinded research analysts (RAs). The treatment groups will be compared with each other at baseline and then at subsequent follow-ups at 3, 6 and 12 months. We will also conduct in-depth, one-to-one interviews with service users from the intervention arm (15-20), carers (15-20) and all therapists involved in the trial. A cost-utility analysis from a healthcare system and societal perspective will be conducted to establish the cost-effectiveness of CaPE against TAU.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients age 18 and above
* Diagnosis of Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) bipolar disorder (both BD I and BD II), currently in remission, confirmed by Structured Clinical Interview for DSM-5 (SCID)
* Currently euthymic (Hamilton Depression Rating Scale, HDRS-17 < 8 and Young Mania Rating Scale, YMRS <8)
* Able to give written informed consent
* On stable psychiatric medication regimen for at least 3 months
* Resident of the trial catchment area.

Exclusion Criteria:

* Active substance use disorder, based on DSM-5 criteria
* Currently experiencing recurrence (mania, hypomania, mixed or depressive
* Active suicidal ideation
* Unstable residential arrangements that reduce likelihood of being available for the duration of trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Interval Follow-up Evaluation | Change in scores from baseline to months 3, 6, and 12
  Longitudinal Interval Follow-up Evaluation (LIFE) is an integrated system for assessing the longitudinal course of psychiatric disorders. The assessment will consist of a semi-structured interview, during which an interviewer uses the LIFE to collect detailed psychosocial, psychopathologic, and treatment information for the follow-up interval. The weekly psychopathology measures are ordinal symptom-based scales with categories defined to match the criteria of the DSM-5.

SECONDARY OUTCOMES:
Demographic Questionnaire | Baseline
  Demographic Questionnaire will be used to assess baseline demographics including age, gender, self-reported sex, marital status, smoking status, employment status, education and monthly income.
Young Mania Rating Scale | Change in scores from baseline to months 3, 6, and 12
  Young Mania Rating Scale (YMRS) will be used to assess manic symptom severity. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours.
Hamilton Depression Rating Scale | Change in scores from baseline to months 3, 6, and 12
  Hamilton Depression Rating Scale (HDRS-17) is a clinician-administered scale that will be used to measure severity of depression symptoms.
Quality of life scale | Change in scores from baseline to months 3, 6, and 12
  EuroQol-5D (EQ- 5D) EQ-5D will be used to assess health-related quality of life over 5 dimensions (mobility, self-care, daily activities, pain-discomfort, anxiety and depression) 44. It also includes and a Visual Analogue Scale that evaluates patients' perceived health status.
Bipolar Recovery Questionnaire | Change in scores from baseline to months 3, 6, and 12
  Bipolar Recovery Questionnaire (BRQ) is a 36-item questionnaire that will be used to measure functioning and personal experiences of recovery specific to patients with BD.
Morisky Medication Adherence Scale-4 items | Change in scores from baseline to months 3, 6, and 12
  Morisky Medication Adherence Scale-4-item will be used to measure medication adherence.
Bipolar Knowledge and Attitudes Questionnaire | Change in scores from baseline to months 3, 6, and 12
  Bipolar Knowledge and Attitudes Questionnaire (BKAQ) is a 25-item questionnaire developed for use in primary care to assess knowledge and attitudes towards bipolar disorder.
Client Service Receipt Inventory | From baseline to months 3, 6, and 12
  Client Service Receipt Inventory (CSRI) is a tool used to collect information on the whole range of services and supports study participants may be accessing.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ishrat Husain, MD, Principal Investigator — Centre for Addiction and Mental Health; Nasim Chaudhry, MD, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Lahore General Hospital, Lahore, Select An Option…, Pakistan

REFERENCES:
- [Derived] Husain MI, Umer M, Asif M, Khoso AB, Kiran T, Ansari M, Aslam H, Bhatia MR, Dogar FA, Husain MO, Khan HA, Mufti AA, Mulsant BH, Naeem F, Naqvi HA, de Oliviera C, Siddiqui MS, Tamizuddin A, Wang W, Zaheer J, Husain N, Chaudhry N, Chaudhry IB. Culturally adapted psychoeducation for bipolar disorder in a low-resource setting: protocol for a multicentre randomised controlled trial. BJPsych Open. 2022 Nov 25;8(6):e206. doi: 10.1192/bjo.2022.598. PMID 36426568